CLINICAL TRIAL: NCT00132509
Title: Comparison of the Classical Rt-PA Procedure (0.9mg/kg Over 60 Minutes) With a Longer Procedure With Lower Dose (0.8mg/kg Over 90 Minutes) in Acute Ischemic Stroke
Brief Title: FRALYSE Trial: Comparison of the Classical Rt-PA Procedure With a Longer Procedure in Acute Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of promotion by the sponsor
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr Paul TROUILLAS, Service de Neurologie, Hôpital Neurologique, Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000.208
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-02

CONDITIONS: Stroke, Acute
Keywords: rt-PA; thrombolysis; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — National Institute of Neurological Disorders and Stroke (U.S.)

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- DFIL (Experimental)
  Interventions: Drug: DFIL
- NINDS (Active Comparator)
  Interventions: Drug: NINDS

INTERVENTIONS:
Drug: DFIL — Alteplase : 0.8mg/kg over 90 minutes
  Arms: DFIL
Drug: NINDS — Alteplase : 0.9mg/kg over 60 minutes
  Arms: NINDS

SUMMARY:
Data from the literature have suggested that a longer time of thrombolysis might be more effective in ischemic stroke. We, the investigators at Hospices Civils de Lyon, have designed a randomized protocol to test this hypothesis. Moreover, the therapeutic window is 7 hours.

Rt-PA (alteplase) is injected intravenously in the 2 arms of the study for a duration of 60 minutes in the arm with a "classical dose" and 90 minutes in the arm with a "low dose-longer infusion".

This is a study of the outcome at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of ischemic stroke
* Presence of a deficit measurable with National Institutes of Health Stroke Scale (NIHSS)
* Lack of any hemorrhagic lesion on the computed tomography (CT) scan at entry
* Time of therapy less than 7 hours after onset of stroke
* Permanent or aggravating symptoms
* Ages 18-81

Exclusion Criteria:

* Lack of cerebral infarction or of cranial trauma within 3 weeks before therapy
* No surgery within 14 days before therapy
* History of cerebral bleeding
* Blood pressure: systolic >185 mmHg and/or diastolic >110 mmHg
* Minor symptoms or symptoms rapidly improving
* Gastro-intestinal or urinary hemorrhage within 21 days
* Arterial puncture within 7 days before therapy
* Epileptic seizure at the beginning of stroke
* Patients under oral anticoagulants or having received heparin within 48 hours, and with elevated activated partial thromboplastin time (aPTT)
* Patients with elevated International Normalized Ratio (INR) or thrombocyte count < 100 x 10^9
* Blood glucose value < 2.7 mmol/l or > 22.2 mmol/l
* Cardiac, pulmonary, hepatic or renal failure, not allowing a study over 3 months
* History of gastric ulcer within 15 days; gestation and menstruation

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2001-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Modified Rankin score | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Paul TROUILLAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Pierre Wertheimer, Bron, France